CLINICAL TRIAL: NCT04408755
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Assessment of the Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AVP-786 program was discontinued, the recruitment was stopped and all participants are no longer being examined or receiving intervention.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-AVP-786-306; 2020-000798-26 (EudraCT Number); 2023-504990-19-00 (EU CTIS Number)
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type
Keywords: Agitation; Dementia of the Alzheimer's type; Alzheimer's disease; AVP-786; Deudextromethorphan hydrobromide; Quinidine sulfate
MeSH Terms: conditions — Psychomotor Agitation; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786 matching placebo capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: Placebo
- AVP-786-18 (Experimental): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-18 (d6-DM 18 milligrams (mg)/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: AVP-786
- AVP-786-42.63 (Experimental): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786 — oral capsules
  Arms: AVP-786-18; AVP-786-42.63
Drug: Placebo — oral capsules
  Arms: Placebo

SUMMARY:
This study was conducted to evaluate the efficacy, safety, and tolerability of AVP-786 (deudextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q]) compared to placebo for the treatment of agitation in participants with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
Eligible participants for this study had a diagnosis of probable Alzheimer's disease (AD) and had clinically significant, moderate/severe agitation secondary to AD.

This was a multicenter, randomized, double-blind, placebo-controlled study, consisting of 12 weeks of treatment. Screening occurred within 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants were randomized into the study.

184 participants were enrolled into the study.

Study medication was administered orally twice daily from Day 1 through Day 85.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of probable Alzheimer's disease according to the 2011 Neuropsychiatric Inventory Agitation/Aggression (NPI-AA) working groups criteria
* Participants with clinically significant, moderate-to-severe agitation for at least 2 weeks prior to Screening that interferes with daily routine per the Investigator's judgment
* Participants who require pharmacotherapy for the treatment of agitation per the Investigator's judgment after an evaluation of reversible factors and a course of nonpharmacological interventions
* Diagnosis of agitation must meet the International Psychogeriatric Association (IPA) provisional definition of agitation.
* Participants meeting an additional predetermined blinded eligibility criterion, which will remain blinded to the clinical study site Investigators and staff
* Participants with a reliable caregiver who is able and willing to comply with all study procedures, including adherence to administering study drug and not administering any prohibited medications during the course of the study, and who spends a minimum of 2 hours per day for 4 days per week with the participant

Exclusion Criteria:

* Participants with dementia predominantly of the non-Alzheimer's type (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia)
* Participants with symptoms of agitation that are not secondary to Alzheimer's dementia (e.g., secondary to pain, other psychiatric disorder, or delirium)
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy [except skin basal-cell carcinoma], poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participants with myasthenia gravis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (45):
  - Clinical Research Site #840-081, Fort Smith, Arkansas
  - Clinical Research Site #840-035, La Jolla, California
  - Clinical Research Site #840-084, Los Angeles, California
  - Clinical Research Site #840-050, Oceanside, California
  - Clinical Research Site #840-064, Pasadena, California
  - Clinical Research Site #840-098, Santa Ana, California
  - Clinical Research Site #840-090, Basalt, Colorado
  - Clinical Research Site #840-009, Atlantis, Florida
  - Clinical Research Site #840-056, Brandon, Florida
  - Clinical Research Site #840-020, Coral Gables, Florida
  - Clinical Research Site #840-059, Doral, Florida
  - Clinical Research Site #840-131, Hialeah, Florida
  - Clinical Research Site #840-039, Jacksonville, Florida
  - Clinical Research Site #840-012, Kissimmee, Florida
  - Clinical Research Site #840-069, Maitland, Florida
  - Clinical Research Site #840-083, Maitland, Florida
  - Clinical Research Site #840-118, Miami, Florida
  - Clinical Research Site #840-004, Miami, Florida
  - Clinical Research Site #840-125, Miami, Florida
  - Clinical Research Site #840-104, Miami, Florida
  - Clinical Research Site #840-133, Miami, Florida
  - Clinical Research Site #840-042, Miami, Florida
  - Clinical Research Site #840-003, Miami, Florida
  - Clinical Research Site #840-036, Orlando, Florida
  - Clinical Research Site 840-111, Pembroke Pines, Florida
  - Clinical Research Site #840-096, Pensacola, Florida
  - Clinical Research Site, Pompano Beach, Florida
  - Clinical Research Site #840-079, Tampa, Florida
  - Clinical Research Site #840-112, Tampa, Florida
  - Clinical Research Site #840-046, Tampa, Florida
  - Clinical Research Site #840-107, West Palm Beach, Florida
  - Clinical Research Site #840-049, Glen Burnie, Maryland
  - Clinical Research Site #840-093, Rochester Hills, Michigan
  - Clinical Research Site #840-015, Hattiesburg, Mississippi
  - Clinical Research Site #840-029, West Long Branch, New Jersey
  - Clinical Research Site #840-072, New Windsor, New York
  - Clinical Research Site #840-097, The Bronx, New York
  - Clinical Research Site #840-095, Monroe, North Carolina
  - Clinical Research Site #840-060, Canton, Ohio
  - Clinical Research Site #840-028, Columbus, Ohio
  - Clinical Research Site #840-061, Edmond, Oklahoma
  - Clinical Research Site #840-099, Tulsa, Oklahoma
  - Clinical Research Site #840-115, McKinney, Texas
  - Clinical Research Site, The Woodlands, Texas
  - Clinical Research Site #840-025, Richmond, Virginia
- Bulgaria (8):
  - Clinical Research Site #100-115, Pernik
  - Clinical Research Site #100-112, Pleven
  - Clinical Research Site #100-106, Plovdiv
  - Clinical Research Site #100-102, Sofia
  - Clinical Research Site #100-111, Sofia
  - Clinical Research Site #100-105, Varna
  - Clinical Research Site #100-108, Varna
  - Clinical Research Site #100-113, Veliko Tarnovo
- Denmark (2):
  - Clinical Research Site # 208-001, Aalborg, North Denmark
  - Clinical Research Site #208-002, Aalborg
- Estonia (3):
  - Clinical Research Site #1 Site #233-002, Tallinn
  - Clinical Research Site #2 Site #233-004, Tallinn
  - Clinical Research Site #233-001, Tartu
- Germany (4):
  - Clinical Research Site #276-017, Böblingen, Baden-Wurttemberg
  - Clinical Research Site #276-005, Bad Homburg, Hesse
  - Clinical Research Site #276-012, Gera, Thuringia
  - Clinical Research Site 276-014, Berlin
- Greece (3):
  - Clinical Research Site# 300-005, Athens
  - Clinical Research Site #300-006, Ioannina
  - Clinical Research Site #300-003, Thessaloniki
- Poland (12):
  - Clinical Research Site #616-018, Zabrze, Katowice
  - Clinical Research Site #616-009, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Clinical Research Site #616-006, Lublin, Lublin Voivodeship
  - Clinical Research Site #616-015, Sochaczew, Masovian Voivodeship
  - Clinical Research Site #616-013, Bydgoszcz
  - Clinical Research Site #616-004, Kielce
  - Clinical Research Site #616-008, Lublin
  - Clinical Research Site #616-010, Lublin
  - Clinical Research Site #616-012, Poznan
  - Clinical Research Site #616-005, Poznan
  - Clinical Research Site #616-001, Pruszcz Gdański
  - Clinical Research Site #616-007, Warsaw
- Portugal (4):
  - Clinical Research Site #620-007, Guimarães, Braga District
  - Clinical Research Site #620-004, Braga
  - Clinical Research Site #620-005, Coimbra
  - Clinical Research Site #620-002, Torres Vedras
- Puerto Rico (4):
  - Clinical Research Site #630-001, Bayamón
  - Clinical Research Site #630-003, Rio Piedras
  - Clinical Research Site #630-002, San Juan
  - Clinical Research Site #630-005, San Juan
- Ukraine (5):
  - Clinical Research Site #804-006, Dnipro
  - Clinical Research Site #804-003, Kharkiv
  - Clinical Research Site #804-004, Kiev
  - Clinical Research Site #804-005, Kyiv
  - Clinical Research Site #804-007, Lviv
- United Kingdom (5):
  - Clinical Research Site #826-003, Blandford Forum
  - Clinical Research Site #826-004, Crowborough
  - Clinical Research Site #826-001, Fulwood
  - Clinical Research Site# 826-006, Manchester
  - Clinical Research Site #826-002, Motherwell

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at clinical sites in the North America and Europe from 13 July 2020 to 27 June 2024.
Pre-assignment Details: A total of 530 participants were screened for the study, of which 184 participants were enrolled and treated with placebo in a 1-week double-blind placebo lead-in period (Period A). A total of 173 participants were then randomized to receive AVP-786 (deudextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q])-18, AVP-786-42.63 or placebo in the 11-week randomization period (Period B).
Groups:
- All Enrolled: Participants received AVP-786 matching placebo capsules, twice a day, for 1 week in Period A.
- AVP-786-18: Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
Period: Period A (Placebo lead-in)
Arm/Group | All Enrolled | Placebo | AVP-786-18 | AVP-786-42.63
Started | 184 | 0 | 0 | 0
Completed | 173 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0
Not completed — Other | 11 | 0 | 0 | 0
Period: Period B (Randomization Period)
Arm/Group | All Enrolled | Placebo | AVP-786-18 | AVP-786-42.63
Started | 0 (173 Participants who completed Period A, were randomized to Period B to receive Placebo, AVP-786-18, and AVP-786-42.63.) | 56 (Out of 173 participants who completed Period A, 56 were randomized to receive matching Placebo.) | 60 (Out of 173 participants who completed Period A, 60 were randomized to receive AVP-786-18 in Period B.) | 57 (Out of 173 participants who completed Period A, 57 were randomized to receive AVP-786-42.63 in Period B.)
Safety Population | 0 | 56 | 60 | 57
Completed | 0 | 44 | 48 | 48
Not Completed | 0 | 12 | 12 | 9
Not completed — Adverse Event | 0 | 3 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0
Not completed — Study Subject Withdrawal by Parent or Guardian | 0 | 2 | 2 | 2
Not completed — Study Terminated by Sponsor | 0 | 1 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 1
Not completed — Reason not Specified | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants who were randomized in the double-blind period B of the study.
Groups:
- Placebo: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786 matching placebo capsules, twice a day, for 11 weeks in Period B.
- AVP-786-18: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
- AVP-786-42.63: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63 | Total
Number analyzed (Participants) | 56 | 60 | 57 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (7.52) | 73.9 (7.85) | 74.8 (6.47) | 75.0 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 42 | 33 | 111
  Male | 20 | 18 | 24 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 5 | 5 | 4 | 14
  White | 50 | 55 | 53 | 158
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 32 | 39 | 36 | 107
  Ethnicity: Not Hispanic or Latino | 22 | 19 | 20 | 61
  Ethnicity: Other | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From the End of Period A (Week 1) to Week 10 in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score
Description: The CMAI is used to assess the frequency of manifestations of agitated behaviors in elderly persons. It consists of 29 agitated behaviors that are further categorized into distinct agitation syndromes, also known as CMAI factors of agitation. These distinct agitation syndromes include aggressive behavior, physically nonaggressive behavior, and verbally agitated behavior. Each of the 29 items is rated on a 7-point scale of frequency (1 = never, 2 = less than once a week but still occurring, 3 = once or twice a week, 4 = several times a week, 5 = once or twice a day, 6 = several times a day, 7 = several times an hour). The ratings are based on the 2 weeks preceding assessment of the CMAI. Higher scores indicate higher frequency of agitated behaviours while lower scores indicate lower frequency of agitated behaviours.
Time Frame: Week 1 to Week 10
Population: Due to discontinuation of development of the AVP-786 compound, no data was collected and analyzed as planned for this pre-specified primary efficacy outcome measure as noted in the SAP. Only safety data was collected and analyzed.
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Serious TEAE
Description: An adverse event (AE) is any untoward medical occurrence or unintended change (eg, physical, psychological, or behavioral), including inter-current illness, that does not necessarily have a causal relationship with the study treatment. A serious adverse event (SAE) is any AE occurring at any dose that results in death, life-threatening experience, persistent or significant disability/incapacity, in-patient hospitalization or prolongation of hospitalization or congenital anomaly/birth defect. TEAEs are all AEs (including serious and non-serious) which started after start of double-blind study drug treatment; or if the event was continuous from baseline and was worsening, serious, study drug related, or resulted in death, discontinuation, interruption or reduction of study therapy.
Time Frame: From randomization (Week 2) up to 30 days after last dose of study drug (Up to Week 16)
Population: Safety population included of all participants who were randomized in the double-blind period B of this study, and took at least one dose of double-blind, randomized study medication. As pre-specified in the Statistical Analysis Plan (SAP), safety data was planned to be collected only for the participants who were randomized in the double-blind period B of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 56 | 60 | 57
Participants
  TEAEs | 20 | 15 | 17
  Serious TEAEs | 1 | 3 | 2

3. Secondary Outcome: Change From the End of Period A (Week 1) to Week 10 in the Clinical Global Impression of Severity of Illness (CGIS) Score, as Related to Agitation
Description: The CGIS is an observer-rated scale that measures illness severity. The CGIS-Agitation is a 7-point (1-7) scale (1 = normal, not at all ill; 7 = among the most extremely ill patients) and assesses severity of agitation in this study. Higher scores indicate severe agitation while the lower scores indicate little or no agitation.
Time Frame: Week 1 to Week 10
Population: Due to discontinuation of development of the AVP-786 compound, no data was collected and analyzed as planned for this pre-specified secondary efficacy outcome measure as noted in the SAP. Only safety data was collected and analyzed.
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization (Week 2) up to 30 days after last dose of study drug (Up to Week 16)
Description: Safety population included of all participants who were randomized in the double-blind period B of this study, and took at least one dose of double-blind, randomized study medication. As pre-specified in the SAP, safety data was planned to be collected only for the participants who were randomized in the double-blind period B of this study.
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
All-Cause Mortality (participants affected / at risk) | 0/56 | 1/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/60 | 2/57
Other Adverse Events (participants affected / at risk) | 20/56 | 14/60 | 17/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | AVP-786-18 (N=60) | AVP-786-42.63 (N=57)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | AVP-786-18 (N=60) | AVP-786-42.63 (N=57)
Idiopathic neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 3
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Mutism (Psychiatric disorders) | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to discontinuation of development of the AVP-786 compound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04408755/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04408755/SAP_001.pdf